CLINICAL TRIAL: NCT03021174
Title: A Feasibility Pilot Study on the Effects of Exercise on Chemotherapy-induced Peripheral Neuropathy and Interoceptive Brain Circuitry
Brief Title: Exercise and Nutrition Interventions During Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ian Kleckner, Research Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RSRB00066046
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Neuropathy;Peripheral
Keywords: CIPN; Chemotherapy-induced peripheral neuropathy
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Exercise for Cancer Patients (EXCAP©®), developed by Dr. Karen Mustian, involves face-to-face instruction and a prescription for an at-home progressive walking and resistance exercise program.
  Interventions: Behavioral: EXCAP Exercise
- Nutrition Education Control (Active Comparator): Nutrition education (control) involves equal time and attention as the exercise arm, but the content covers nutrition for cancer patients and lacks an exercise prescription.
  Interventions: Behavioral: Nutrition Education Control

INTERVENTIONS:
Behavioral: EXCAP Exercise — 12 weeks of at-home walking and resistance exercise
  Arms: Exercise
Behavioral: Nutrition Education Control — 12 weeks of implementing eating tips
  Arms: Nutrition Education Control

SUMMARY:
This is a feasibility pilot study to initiate a research program to assess the effects of exercise on chemotherapy-induced peripheral neuropathy (numbness, tingling, and pain in the hands and feet).

DETAILED DESCRIPTION:
This is a feasibility pilot study to help obtain external funding for a larger study to assess the effects of exercise on chemotherapy-induced peripheral neuropathy (CIPN), which is a dose-limiting and painful side effect of chemotherapy for which there are no established treatments. The investigators will conduct a two-arm randomized clinical trial in 40 cancer patients receiving chemotherapy where Arm 1 is 12 weeks of exercise during chemotherapy and Arm 2 is 12 weeks of nutrition education (control condition) during chemotherapy. The investigators will acquire data on CIPN via patient reports and clinical assessments as well as general pain and hypothetical mechanistic factors that may help explain how exercise may treat CIPN; these factors include measures of musculoskeletal, cardiovascular, neuropsychological, and immunological function. The primary outcomes are related to the feasibility of identifying, recruiting, and obtaining complete data from research participants.

ELIGIBILITY:
Inclusion Criteria:

* Have non-metastatic cancer
* Be chemotherapy naïve
* Be scheduled to receive CIPN-inducing chemotherapy during the study (platinums, vinca alkaloids, taxanes, thalidomide, or bortezomib) for the duration of the intervention (12 weeks)
* Report symptoms of peripheral neuropathy at baseline (subject-reported severity of numbness and tingling in hands/feet of at least 1 on a 0-10 scale)
* Be able to perform the exercise intervention
* Be able to read English
* Be at least 18 years old (no upper limit on age)
* Be consistently right-handed in daily activities for consistency in reporting any lateralized effects from brain imaging
* Provide written informed consent

Exclusion Criteria:

* Receive surgery, radiation, or hormone therapy for their cancer during the study
* Be in the active or maintenance stage of exercise behavior (i.e., subjects must be sedentary)
* Have contraindications for MRI scanning (pacemaker, metal implants, pregnancy, etc. - note that most port-a-caths are safe for MRI scanning)
* Have physical limitations (e.g., cardiorespiratory, orthopedic, central nervous system) that contraindicate participation in maximal physiological fitness testing and a low/moderate intensity home-based walking and progressive resistance exercise program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
Percent of patients screened who are eligible | 12 weeks
  Number of patients eligible divided by number of patients screened
Percent of patients eligible who are consented | 12 weeks
  Number of patients consented divided by number of patients approached
Percent of patients consented who complete the exercise intervention | 12 weeks
  Number of patients in exercise arm who improve daily steps divided by number of patients in exercise arm
Percent of patients consented who complete pre- and post-intervention measures of the patient-reported assessment of chemotherapy-induced peripheral neuropathy | 12 weeks
  Number of patients who completed pre- and post-intervention CIPN-20 questionnaire divided by number of patients consented (both arms)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No
Interested researchers may contact the study PI with requests for collaboration.

REFERENCES:
- [Derived] Kleckner IR, Manuweera T, Lin PJ, Chung KH, Kleckner AS, Gewandter JS, Culakova E, Tivarus ME, Dunne RF, Loh KP, Mohile NA, Kesler SR, Mustian KM. Pilot trial testing the effects of exercise on chemotherapy-induced peripheral neurotoxicity (CIPN) and the interoceptive brain system. Support Care Cancer. 2024 Sep 21;32(10):677. doi: 10.1007/s00520-024-08855-y. PMID 39304604
- [Derived] Kleckner IR, Manuweera T, Lin PJ, Chung KH, Kleckner AS, Gewandter JS, Culakova E, Tivarus ME, Dunne RF, Loh KP, Mohile NA, Kesler SR, Mustian KM. Pilot trial testing the effects of exercise on chemotherapy-induced peripheral neurotoxicity (CIPN) and the interoceptive brain system. Res Sq [Preprint]. 2024 Mar 13:rs.3.rs-4022351. doi: 10.21203/rs.3.rs-4022351/v1. PMID 38559210